CLINICAL TRIAL: NCT07273851
Title: A Randomized Controlled Trial Comparing Propofol and Ketofol for Hemodynamic Stability During Electroconvulsive Therapy
Brief Title: Comparison of Propofol and Ketofol as Induction Agents for Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fauji Foundation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFH-PropKet-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: Propofol Ketofol Electroconvulsive Therapy Anesthesia Hemodynamic Stability
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Participants receive intravenous propofol (1 mg/kg) as the induction agent for modified electroconvulsive therapy (ECT). Glycopyrrolate (0.004 mg/kg) is given as premedication, and Ringer's lactate is started before induction. ECT is performed using bifrontotemporal electrodes under standard monitoring. Systolic blood pressure is recorded 20 minutes after shock delivery.
  Interventions: Drug: Propofol
- Ketofol group (Active Comparator): Participants receive ketofol (a 1:1 mixture of ketamine and propofol) as the induction agent for modified ECT. Ketofol is prepared by mixing propofol 0.5 mg/kg and ketamine 0.5 mg/kg in the same syringe. Standard premedication and monitoring apply. Systolic blood pressure is recorded 20 minutes after shock delivery.
  Interventions: Drug: Ketofol

INTERVENTIONS:
Drug: Propofol — Intravenous induction agent administered before electroconvulsive therapy. Participants in this arm will receive IV propofol 1 mg/kg as a single slow bolus immediately before ECT under continuous ECG, pulse oximetry, and non-invasive blood pressure monitoring. Premedication with glycopyrrolate 0.004 mg/kg IV will be given to all patients. Ringer's lactate infusion will begin prior to induction. After loss of eyelash reflex, ECT will be performed using bifrontotemporal electrodes. Systolic blood pressure, heart rate, and oxygen saturation will be recorded at baseline and 20 minutes after shock delivery. The patient will be ventilated with 100 % oxygen until spontaneous breathing resumes.
  Arms: Propofol group
Drug: Ketofol — Intravenous admixture prepared immediately before induction by combining equal parts of ketamine and propofol in the same syringe. Participants will receive propofol 0.5 mg/kg + ketamine 0.5 mg/kg as a slow IV bolus immediately before ECT. Continuous ECG, pulse oximetry, and non-invasive blood pressure monitoring will be maintained. Premedication and procedural steps are identical to the propofol arm. The rationale is that ketamine's sympathetic stimulation counterbalances the hypotensive effect of propofol, potentially improving hemodynamic stability during ECT. Hemodynamic variables and seizure duration will be documented at baseline, during, and 20 minutes after shock delivery. Patients will receive 100 % oxygen ventilation until spontaneous respiration resumes.
  Arms: Ketofol group

SUMMARY:
This randomized controlled trial will compare two anesthetic agents, propofol and ketofol (a combination of propofol and ketamine), in patients undergoing electroconvulsive therapy (ECT). Propofol is commonly used but may lower blood pressure, while ketofol may help maintain more stable cardiovascular function. The study will evaluate changes in systolic blood pressure following ECT when either propofol or ketofol is used for anesthesia induction. A total of 80 adult patients will be enrolled and randomly assigned to one of the two treatment groups. Findings may guide anesthesiologists in selecting the safest and most effective induction agent for ECT.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is an established treatment for depression and other psychiatric disorders that do not respond to medications. The procedure requires short-term anesthesia. Propofol is the most commonly used drug for anesthesia during ECT because it acts quickly and allows patients to recover rapidly, but it is often linked with low blood pressure and shorter seizure duration. Ketamine, another anesthetic drug, increases blood pressure and heart rate and may prolong seizures, but it is rarely used alone because of side effects such as agitation.

A newer approach is to combine both drugs, known as ketofol, to balance their effects. This study will directly compare propofol and ketofol as induction agents during ECT, with a focus on how each affects systolic blood pressure. Eighty adult patients scheduled for ECT will be randomly assigned to receive either propofol or ketofol for anesthesia. Blood pressure will be measured before and after the procedure, and additional information such as seizure duration, recovery time, and side effects will be recorded. The results will provide evidence on whether ketofol offers better hemodynamic stability than propofol alone, potentially improving safety during ECT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years

Both genders

ASA physical status I-II

Scheduled for electroconvulsive therapy

Exclusion Criteria:

* History of chronic opioid therapy

Pregnancy

Known allergy or hypersensitivity to propofol or ketamine

History of cardiovascular disease

History of renal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Mean Systolic Blood Pressure 20 Minutes After Electroconvulsive Therapy | 20 minutes after seizure stimulus during the index ECT session
  Systolic blood pressure (SBP) will be recorded 20 minutes after the delivery of electrical stimulus in both study groups using a non-invasive blood pressure monitor. Baseline SBP will also be recorded prior to induction. The mean SBP between propofol and ketofol groups will be compared to determine the effect of anesthetic agent on post-ECT hemodynamic stability.

SECONDARY OUTCOMES:
Heart Rate at 20 Minutes Post-ECT | 20 minutes post-ECT
  Heart rate will be measured at baseline, immediately after ECT, and 20 minutes post-shock to compare cardiovascular response between the two groups.
Seizure Duration | Immediately following ECT
  Duration of the ECT-induced seizure will be measured in seconds using EEG tracing or motor observation from the time of electrical stimulus until cessation of seizure activity.
Recovery Time | Up to 30 minutes after ECT
  Time in minutes from the completion of ECT to spontaneous respiration and recovery of consciousness (Aldrete score ≥ 9) will be recorded to assess recovery profile.
Incidence of Hypotension | From induction until 30 minutes post-ECT
  The occurrence of hypotension (defined as a ≥20% decrease from baseline mean arterial pressure) during or after ECT will be documented and compared between groups.
Oxygen Saturation (SpO₂) | Baseline, intra-procedure, and up to 30 minutes post-ECT
  Minimum oxygen saturation will be monitored continuously using pulse oximetry and recorded to identify any desaturation episodes during and after ECT.
Adverse Events | Intraoperative period and recovery up to 30 minutes post-ECT
  Any adverse event such as nausea, vomiting, arrhythmia, emergence agitation, or hallucination will be recorded and compared between the two study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Fauji Foundation Hospital, Rawalpindi, Pakistan, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikiz C, Gunenc F, Iyilikci L, Ozbilgin S, Ellidokuz H, Cimilli C, Mermi Z, Gokel E. Effects of Propofol and Propofol-Remifentanil Combinations on Haemodynamics, Seizure Duration and Recovery during Electroconvulsive Therapy. Turk J Anaesthesiol Reanim. 2021 Feb;49(1):44-51. doi: 10.5152/TJAR.2020.157. Epub 2020 Dec 16. PMID 33718905
- [Background] Mehta D, Palta S, Gupta N, Saroa R. Comparison of effect of etomidate with propofol on hemodynamics during modified electroconvulsive therapy. J Anaesthesiol Clin Pharmacol. 2022 Jan-Mar;38(1):104-110. doi: 10.4103/joacp.JOACP_185_20. Epub 2022 Apr 25. PMID 35706636
- [Background] Guha D, Sheshadri K, Singh S, Bhan S. Efficacy of propofol versus ketamine in modified electroconvulsive therapy: a prospective randomized control trial. J Acute Dis. 2022;11(3):89-93.
- [Background] Smischney NJ, Beach ML, Loftus RW, Dodds TM, Koff MD. Ketamine/propofol admixture (ketofol) is associated with improved hemodynamics as an induction agent: a randomized, controlled trial. J Trauma Acute Care Surg. 2012 Jul;73(1):94-101. doi: 10.1097/TA.0b013e318250cdb8. PMID 22743378
- [Background] Smischney NJ, Seisa MO, Morrow AS, Ponce OJ, Wang Z, Alzuabi M, Heise KJ, Murad MH. Effect of Ketamine/Propofol Admixture on Peri-Induction Hemodynamics: A Systematic Review and Meta-Analysis. Anesthesiol Res Pract. 2020 May 8;2020:9637412. doi: 10.1155/2020/9637412. eCollection 2020. PMID 32454816